CLINICAL TRIAL: NCT05982535
Title: The Application of Neopep-S Ingredient Easy Dew MD Regen Cream in the Indication of Dry Skin A Prospective Researcher-led Clinical Study to Assess Efficacy and Safety
Brief Title: Neopep-S Ingredient Easy Dew MD Regen Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eun-ji Kim (Industry)
Responsible Party: Sponsor-Investigator, Eun-ji Kim, Clinical Trial Manager, CGBio Inc.
Organization: CGBio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G2206
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Dry Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Easy Dew MD Regen Cream (Experimental): The subject applies the provided medical device twice a day (morning and evening) to areas with symptoms of dry skin so that it can be absorbed well.
  Interventions: Device: Easy Dew MD Regen Cream
- Physiogel Stability Intensive Cream MD (Active Comparator): The subject applies the provided medical device twice a day (morning and evening) to areas with symptoms of dry skin so that it can be absorbed well.
  Interventions: Device: Easy Dew MD Regen Cream

INTERVENTIONS:
Device: Easy Dew MD Regen Cream — The subject applies the provided medical device twice a day (morning and evening) to areas with symptoms of dry skin so that it can be absorbed well.
  Other Names: Physiogel Stability Intensive Cream MD

SUMMARY:
The purpose of this clinical study is to provide patients diagnosed with dry skin due to various causes such as atopic dermatitis and Yangjin The effect on skin regeneration after applying EasyDew MD Regen Cream containing Neopep-S, a regeneration factor, and It is intended to assess safety.

DETAILED DESCRIPTION:
The total study period for this clinical study is 12 months from the date of IRB approval, led by researchers from a single institution It's a clinical study. The individual participation period of the participant is one month.

Subjects are those diagnosed with dry skin due to a variety of factors (and/or courts) Agents) perform screening tests after agreeing in writing to participate in the clinical study.

Evaluating the screening test results, and subjects who meet the selection criteria and do not meet the exclusion criteria, for clinical research It must be registered. Random assignments of the study group and control group are conducted in a random number table at a 5:5 ratio.

* Control group: 10 people with dexian med cream
* Research Group: 10 people applying EasyDew MD Regen Cream Clinical study subjects are randomly assigned to control and study groups. The control group is Dexian, a foreign medical device product Med cream is applied, and in the case of the study group, EasyDewMD Regen cream provided through prescription is applied. clinical practice Subjects apply an appropriate amount twice a day (morning and evening) to skin areas with dry skin symptoms and can be absorbed well Let's make it happen. After applying the medical device for clinical research, the progress is observed for one month, and the subject is subject to about one month of clinical research During the period, research institutes will be regularly visited to evaluate their validity and safety on the day of screening (Visit1), the day of medical device application (Visit2), 2 weeks after medical device application (Visit3), and 1 month after application (Visit4).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with xerotic skin among adults aged 19 to 80 years
2. Subjects who have voluntarily decided to participate in this clinical study and signed a written informed consent

Exclusion Criteria:

1. Subjects with uncontrolled diabetes
2. Immunosuppressants, corticosteroids, cytotoxic drugs, anticoagulants, etc. are included in the results You are on long-term or scheduled to receive medication that may affect you a person who is subject to
3. Acute or chronic skin disease; stage in progress or active in the area of application Subject to bacterial or viral infection
4. Where the researcher's judgment determines that participation in the study is inappropriate

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss | before and one month after medical device application
  Percutaneous moisture loss measured

SECONDARY OUTCOMES:
Investigator Global Assessment Scale | before medical device application and one month after medical device application
  Assess the patient's overall condition /lowest 0 score ( best score) to highest 30 score( worst score)
Dermatology Life Quality Index | before medical device application and one month after medical device application
  Assess patient quality of life / lowest 0 score ( best score) to highest 4 score( worst score)
Itching score | before medical device application and one month after medical device application
  Evaluate the Itching scale / lowest 1 score ( best score) to highest 5 score( worst score)

CONTACTS AND LOCATIONS:
Overall Officials: Jihye Lee, Study Director — CGBio Inc.
Locations (1):
- Ajou University Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No